CLINICAL TRIAL: NCT02049723
Title: How Much do Patients With Gastroesophageal Disease Know About Their Own Disease in Korea?
Brief Title: Assessment of GERD Knowledge Level Among Patients With it in Korea
Acronym: GERD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Yeonsoo Kim, Assistant professor, Chuncheon Sacred Heart Hospital
Other Study IDs: GERDclub2013-97
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Esophagitis, Reflux
Keywords: Gastroesophageal reflux disease; Knowledge
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with GERD: The knowledge level on GERD among Korean patients with gastroesophageal disease was evaluated by the method of multicenter survey

SUMMARY:
* 1. Research topic: How much do patients with GERD know about their own disease in Korea? (multicenter survey)
* 2. Questionnaires for multicenter survey:

  1. Questionnaire 1 - include items for basic characteristics of participant patients
  2. Questionnaire 2 - modification of GERD knowledge test which was used in BMC Health Services Research 2008;8:236 (Prof. Jorgen Urnes)
* 3. Subjects: patients with GERD in secondary or tertiary hospital
* 4. Participant institutes: GERD club members, The Korean Society of Neurogastroenterology and Motility

DETAILED DESCRIPTION:
Validation process to produce Korean version of GERD knowledge test

1. Forward Translation of GERD knowledge test of prof. Jorgen Urnes: through certified translation company
2. Expert's review of the forward translated knowledge test : among members of GERD club,
3. Pilot survey among nurses and some patients
4. Korean Version, provisional
5. Backward translation: through certified translation company
6. Consultation with Prof. Jorgen Urnes about backward translated knowledge test
7. Korean Version, final
8. Print and distribution
9. Study start

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as GERD by doctors

Exclusion Criteria:

* Patients without GERD

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GERD who visit the secondary or tertiary University hospital for their treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Proportion (%) of patients with GERD who seek more information on GERD which represents the necessity of effective educational programs on the disease in Korea | 1 year
  GERD. gastroesophageal reflux disease

SECONDARY OUTCOMES:
Average score in GERD knowledge test which means GERD knowledge level of the patients | 1 year
  GERD, gastroesophageal reflux disease

CONTACTS AND LOCATIONS:
Overall Officials: Moo In Park, MD, Study Director — Professor, Department of Internal Medicine, Kosin University Gospel Hsopital
Locations (1):
- Yeon-Soo Kim, Chuncheon, Gangwon-do, South Korea